CLINICAL TRIAL: NCT07220798
Title: Improving Self-Care of Caregivers of Adults in Homecare With Heart Failure and Cognitive Impairment (ViCCY)
Brief Title: Virtual Caregiver Coach for You (ViCCY)
Acronym: ViCCY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Visiting Nurse Service of New York (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1R01AG094822 (NIH)
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Cognitive Impairment; Caregiver Burden
Keywords: heart failure; cognitive impairment; caregiver burden; caregiver stress; self-care; dyads
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: This study is based on both the Transactional Model of Stress and Coping and the Dyadic Health Behavior Change model. The stressor for caregivers is the demand of caregiving. This stressor commonly causes stress in the relationship. The response to this stressor is influenced by appraisal of the stress, resources, problem management, and support resources, factors used in the ViCCY intervention. In patients, caregiver stress, combined with the stress of illness, accentuates cognitive, affective, and somatic symptoms, thereby impairing mental health. Interdependence is captured in the Dyadic Health Behavior Change model, which emphasizes the individual contributions of both the patient and the caregiver while simultaneously recognizing the synergy of the relationship.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and all staff involved in collecting assessment data will be blinded to group assignment until after the data are locked. The coach providing the intervention, Dr. Hirschman (fidelity), and the caregiver participants will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ViCCY Intervention (Experimental): The intervention group will receive 10 sessions of ViCCY over 6-months.
  Interventions: Behavioral: ViCCY
- Usual Care (No Intervention): Usual Home Health Care.

INTERVENTIONS:
Behavioral: ViCCY — The intervention group will receive 10 Health Coach sessions of ViCCY over 6-months.
  Arms: ViCCY Intervention

SUMMARY:
This RCT design will enroll 254 informal caregivers (spouse/partner or child) of HHC patients with HF/CI and 60 patients with HF and mild to moderate CI (60 dyads). After collecting baseline data, we will block randomize the caregivers 1:1 to the ViCCY intervention or comparator group, stratifying randomization by caregiver sex (male/female), relationship (spouse/partner or child), and race (white/other)- factors known to influence caregiving burden, perceived stress, and receptivity to the intervention. We will encourage caregivers to use their own devices but provide tablet devices with wireless network access if needed. The intervention group will receive 10 sessions of ViCCY over 6 months.

DETAILED DESCRIPTION:
Purpose and Specific Aims

Cognitive Impairment (CI) has been reported to be as high as 78% in older adults with Heart Failure (HF). CI markedly increases the risk of adverse HF outcomes such as hospitalization and death, and patients with CI and HF are rarely able to manage without a caregiver. The high level of caregiving demands lead to an increase in stress and strained relationships with caregiving recipients, which can lead to poor coping and decreased mental health among caregivers. This study aims to test a self-care intervention (Virtual Caregiver Coach for You -ViCCY) targeting caregivers to support mental health and explore whether changes in caregiver mental health impacts patient outcomes. We will examine relationship strain as the primary mechanism for improvements in outcomes in patients and caregivers.

Aim 1: Test the efficacy of ViCCY vs. UC in improving outcomes of caregivers of home health care (HHC) patients with HF/CI.

Aim 2: Explore the effect of ViCCY on outcomes in HHC patients with HF/CI. At 6-months we will report differences in mental health measured with the SF-36 and its contributors of depression, anxiety, and somatic HF symptoms between patients whose caregivers are randomized to ViCCY compared to UC.

Aim 3: Describe the mechanisms by which outcomes are achieved.

Overview of Study Design and Methods

This RCT design will enroll 254 informal caregivers (spouse/partner or child) of HHC patients with HF/CI and 60 patients with HF and mild to moderate CI (60 dyads). After collecting baseline data, we will block randomize the caregivers 1:1 to the ViCCY intervention or comparator group, stratifying randomization by caregiver sex (male/female), relationship (spouse/partner or child), and race (white/other)- factors known to influence caregiving burden, perceived stress, and receptivity to the intervention. We will encourage caregivers to use their own devices but provide tablet devices with wireless network access if needed. The intervention group will receive 10 sessions of ViCCY over 6 months.

Participant Recruitment and Data Collection

Participants will be (254) caregivers of community dwelling older adults with HF/CI and 60 dyads (caregivers and patients) with HF and mild to moderate CI.

Data Sources and Analysis

We will use an intent-to-treat approach with the primary outcomes assessed at baseline, 3- and 6-months, and 12-months. Efficacy will be analyzed at 6-months. We will summarize participant characteristics using descriptive statistics. Shapiro-Wilk and Levin's tests will be used to assess distributional assumptions of normality. Mixed effects regression models will be used to assess intervention efficacy. Outcomes will be assessed using pre-post self-reported survey data.

ELIGIBILITY:
Inclusion Criteria:

* Patient Inclusion Criteria

  1. Older adults (=>50 years of age)
  2. Enrolled in Home Health Care
  3. Documented to have HF
  4. Mild to moderate CI on the BIMS or OASIS items
  5. Able to provide informed consent
  6. Able to provide self-report data
* Caregiver Inclusion Criteria

  1. Adults (=>18 years of age)
  2. Spouse/partner or child living with or in close proximity to the patient
  3. Caregiver of a home care patient who is currently receiving or recently received services and who has mild to severe cognitive impairment
  4. Reporting poor self-care on screening (Health Self-Care Neglect scale score =>2)
  5. Reporting poor mental health on screening (screened with the PROMIS Global Mental Health 4a score <12)
  6. Caregiving or supporting the patient at least 8 hours/week
  7. Able to complete the protocol, e.g., adequate vision and hearing, English speaking.
  8. Able to provide informed consent
  9. Able to use technology

Exclusion Criteria:

* Patient Exclusion Criteria

  1. Dementia (ICD-10 code for dementia)
  2. Enrolled in hospice
  3. Non-English speaking
* Caregiver Exclusion Criteria 1. Non-English speaking

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2028-06-14 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Short Form Health Survey (SF-36) (Both) | Baseline, 3- and 6- and 12-months
  Mental health is a state of mental well-being that enables people to cope with the stresses of life, realize their abilities, learn well and work well. The SF-36 provides standardized scores and national norms for comparison. The SF-36 is valid in many populations and caregivers. It is one of the common data elements.

SECONDARY OUTCOMES:
Self-Care of Informal Caregiver Inventory (Caregiver) | Baseline, 3- and 6- and 12-months
  Behaviors performed to maintain health
Perceived Stress Scale short form (Caregiver) | Baseline, 3- and 6- and 12-months
  Demands exceed ability to cope
Brief-COPE (Caregiver) | Baseline, 3- and 6- and 12-months
  Ability to respond to stressors with appropriate adaptive coping resources.
Dyadic Relationship Scale (Both) | Baseline, 3- and 6- and 12-months
  Measure of strain in the dyadic relationship
HF Caregiver Questionnaire (Patient) | Baseline, 3- and 6- and 12-months
  load experienced when caring for a loved one
Patient Health Questionnaire (PHQ-9) (Patient) | Baseline and 6-months
  Measures signs and symptoms of depression.
Generalized Anxiety Disorder (GAD-7) (Patient) | Baseline and 6-months
  Measures signs and symptoms of Anxiety.
HF Somatic Perception Scale (Patient) | Baseline and 6-months
  Measures symptoms of Heart Failure.
Charlson Comorbidity Index (Patient) | Baseline and 6-months.
  Captures patient Medications and Chronic Conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Riegel, PhD, RN, Principal Investigator — VNS Health (formerly Visiting Nurse Service of New York)

IPD SHARING:
Plan to Share IPD: No